CLINICAL TRIAL: NCT01101230
Title: Effects of a Diet Rich in Almonds on LDL Cholesterol, LDL Particle Size, Abdominal Adiposity and Vascular Health
Brief Title: Effects of Almonds on Cardiovascular Risk Factors
Acronym: ALD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PKE 104
Record Dates: First submitted 2010-03-24; First posted 2010-04-09 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; cholesterol; low-density; lipoprotein; high-density lipoprotein; triglycerides
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Almond (Experimental)
  Interventions: Other: Almonds
- Muffin (Placebo Comparator)
  Interventions: Other: Almonds

INTERVENTIONS:
Other: Almonds — 1.5 oz almonds/day

SUMMARY:
The purpose of this research is to build the evidence base for approval of FDA health claims related to almonds and cardiovascular disease. A randomized, 2-period, crossover controlled feeding study was designed to compare the effects of two blood cholesterol lowering diets that meet the American Heart Association recommendations. The nutrient profiles of the control diet (no almonds/day) and almond diet (1.5 oz. of almonds/day) are matched for protein, saturated fat, and cholesterol. The study population consists of two cohorts of 25 men and women with moderately elevated LDL-C. The investigators hypothesize that a cholesterol-lowering diet designed with almonds confers greater cardioprotective effects than a cholesterol-lowering diet without almonds on the basis of the LDL-C lowering response, effect on LDL particle size, abdominal adiposity and vascular health.

ELIGIBILITY:
Inclusion Criteria:

* BMI (20-35)
* Low density lipoprotein cholesterol males (128-194mg/dL) and females (121-190 mg/dL)

Exclusion Criteria:

* Pregnant, planning to become pregnant, or lactating
* Smoking; cholesterol-lowering medication
* Glucose-lowering medication
* Over the counter cholesterol-lowering substances (e.g.: psyllium, fish oil, soy lecithin, phytoestrogen)
* The following medical conditions:

  * heart disease
  * stroke
  * Heart attack
  * blood pressure >140/90
  * diabetes
  * renal or kidney disease
  * rheumatoid arthritis
  * blood clotting disorder
  * liver disease or cirrhosis
  * compromised immune system
  * peripheral vascular disease or circulation problems

    *> 10% body weight loss in the past 6 months
  * vegetarian
  * nut allergies

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Lipid/lipoprotein profile | End of diet period 1 (week 6) and diet period 2 (week 14)
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides are measured as part of the lipoprotein profile.
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).

SECONDARY OUTCOMES:
Additional lipid/lipoprotein measures (VLDL, IDL, and remnant lipoproteins) | End of diet period 1 (week 6) and diet period 2 (week 14)
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).
Lipoprotein (LDL, HDL, VLDL, IDL) subclasses | End of diet period 1 (week 6) and diet period 2 (week 14)
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).
Abdominal adiposity as measured by dual-energy x-ray absorptiometry | End of diet period 1 (week 6) and diet period 2 (week 14)
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).
Leg adiposity as measured by dual-energy x-ray absorptiometry | End of diet period 1 (week 6) and diet period 2 (week 14)
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).
Apolipoproteins (A1 and B) | End of diet period 1 (week 6) and diet period 2 (week 14)
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).
Vascular health (plasma nitric oxide) | End of diet period 1 (week 6) and diet period 2 (week 14)
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).
Total body composition as measured by dual-energy x-ray absorptiometry | End of diet period 1 (week 6) and diet period 2 (week 14)
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).
Waist circumference | End of diet period 1 (week 6) and diet period 2 (week 14)
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).
HDL functionality (cholesterol efflux) | End of diet period 1 (week 6) and diet period 2 (week 14)
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).
Cholesterol absorption/synthesis (measured by plasma plant sterols and cholesterol precursors) | End of diet period 1 (week 6) and diet period 2 (week 14)
  Diet period one runs for 6 weeks, then there is a 2 week compliance break, and then diet period two runs for 6 weeks (total time commitment is 14 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, Principal Investigator — Penn State University; Claire E Berryman, Study Director — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Berryman CE, Fleming JA, Kris-Etherton PM. Inclusion of Almonds in a Cholesterol-Lowering Diet Improves Plasma HDL Subspecies and Cholesterol Efflux to Serum in Normal-Weight Individuals with Elevated LDL Cholesterol. J Nutr. 2017 Aug;147(8):1517-1523. doi: 10.3945/jn.116.245126. Epub 2017 Jun 14. PMID 28615375
- [Derived] Berryman CE, West SG, Fleming JA, Bordi PL, Kris-Etherton PM. Effects of daily almond consumption on cardiometabolic risk and abdominal adiposity in healthy adults with elevated LDL-cholesterol: a randomized controlled trial. J Am Heart Assoc. 2015 Jan 5;4(1):e000993. doi: 10.1161/JAHA.114.000993. PMID 25559009